CLINICAL TRIAL: NCT04385433
Title: A Comparative Study of Pravastatin vs Placebo as Primary Prevention of Severe Subcutaneous Breast Fibrosis in Hyper-radiosensitive Identified Patients With Breast Cancer
Acronym: PRAVAPREV-01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough patients enrolled
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROICM 2019-11 PRA
Record Dates: First submitted 2020-04-23; First posted 2020-05-13 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): RADIOTHERAPY + PRAVASTATIN
  Interventions: Drug: EXPERIMENTAL ARM; Radiation: Standard adjuvant whole breast radiotherapy (50Gy/ 25 fractions to whole breast) followed or not by a boost to tumor bed (16Gy/ 8 fractions)
- CONTROL GROUP (Placebo Comparator): RADIOTHERAPY + PLACEBO
  Interventions: Other: CONTROL GROUP; Radiation: Standard adjuvant whole breast radiotherapy (50Gy/ 25 fractions to whole breast) followed or not by a boost to tumor bed (16Gy/ 8 fractions)

INTERVENTIONS:
Drug: EXPERIMENTAL ARM — Patients in the experimental arm will receive:
  * Daily pravastatin (40mg/d) during 12 months (pravastatin initiation: first day of radiotherapy).
  * Standard adjuvant whole breast radiotherapy (50Gy/ 25 fractions to whole breast) followed or not by a boost to tumor bed (16Gy/ 8 fractions).
  Other Names: pravastatin group
  Arms: EXPERIMENTAL GROUP
Other: CONTROL GROUP — Patients in the standard arm will receive:
  * Daily placebo during 12 months (placebo initiation: first day of radiotherapy)
  * Standard adjuvant whole breast radiotherapy (50Gy/ 25 fractions to whole breast) followed or not by a boost to tumor bed (16Gy/ 8 fractions).
  Other Names: placebo group
  Arms: CONTROL GROUP
Radiation: Standard adjuvant whole breast radiotherapy (50Gy/ 25 fractions to whole breast) followed or not by a boost to tumor bed (16Gy/ 8 fractions) — Radiotherapy will last 5 weeks during treatment by Pravastatine or Placebo

SUMMARY:
-Interventional trials aim at preventing severe RIF occurrence in BC patients selected by individual radiosensitivity:

PRAVAPREV-01 will be the first interventional double blind trial that will offer a personalised strategy to breast cancer patients who will be treated with adjuvant RT after breast conserving surgery:

* By assessing individual risk of severe RIF development
* By offering a statin targeted therapy to the high-risk patients identified.

DETAILED DESCRIPTION:
According to VICAN5 report, near 50% of survivorship breast cancer (BC) patients suffered impairment of their QoL 2 and 5 years after BC diagnosis compared to overall population. In France, adjuvant radiotherapy (RT) is performed to 88.5% of BC patients. Severe toxicities after adjuvant RT such as radio-induced fibrosis (RIF) in BC patients can have a negative impact on quality of life and a marked effect on subsequent psychological outcomes.

However, current practice standards commonly prescribe RT irrespective of the individual radiosensitivity risk. This study propose to identify BC at high RIF risk and to prevent severe RIF occurrence in this selected BC population by the use of anti-fibrotic agent (pravastatin).

How to identify the risk of individual radiosensitivity? Since 1995 a rapid (72 h) radiosensitivity assay based on flow cytometric assessment of radiation-induced CD8 T-lymphocyte apoptosis (RILA) has been developed. A lot of laboratory observed a significant relationship between RILA and toxicities occurrence, in particular in a prospective multicenter French study (NCT00893035, Azria et al, EBioMedicine 2015). Data from this study have validated the use of the NovaGray RILA Breast® test in clinical routine and enabled its CE-mark obtention in 2016.

How to prevent severe RIF occurrence? Few phase II clinical trials have assessed anti-fibrotic properties of some drugs in a preventive setting (pentoxyfilline/vitamine E, ambroxol, ACE inhibitors, amifostine) and showed controversial results regarding efficacy and/ or tolerance. To date, no large phase III clinical trial confirmed these therapeutic strategies in the prevention of severe breast RIF occurrence.

Since 2000, Rho/ROCK pathway inhibition habe been showed, in particular by Pravastatin, was able to prevent and cure severe RIF in different preclinical RIF models. Based on those results, a phase II clinical trial PRAVACUR (NCT01268202) has been conducted,assessing efficacy of 12-months daily pravastatin delivered in patients with established RIF after head and neck radiotherapy. The use of Pravastatin significantly reduced RIF grade in 51% of patients (clinical assessment at 12-months) without any rebound effect after pravastatin completion (Bourgier IJROBP 2019).

This hypothesis is therefore that pravastatin given in a preventive approach will significantly decrease severe breast fibrosis occurrence in a highly selected breast cancer population treated by adjuvant breast RT and considered at high risk of RIF (tailored by the NovaGray RILA Breast® test).

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years old (no age limit)
2. Conservative breast cancer surgery
3. High risk level of breast fibrosis identified by the centralized NovaGray RILA Breast® test
4. Invasive carcinoma : pT1-T2; pN0 (negative sentinel nodes or axillary nodes dissection) and/or Ductal in situ carcinoma
5. Negative surgical margins
6. Indication of whole breast irradiation only (with or without boost to tumor bed according to physician discretion)
7. Only 3D-conformal RT will be allowed
8. Blood sample allowing pravastatin use : serum creatinine ≤ 130 µmol/l; ASAT and ALAT≤ 2N; total bilirubin ≤ 1.5N; CK MM levels < 3 x ULN for women ≥ 70 years (at least 15 days before randomization).
9. Negative pregnancy test in women of childbearing potential (β-HCG dosage ≤ 7 days prior to randomization), an adequate contraception should be used from the beginning of the study to 4 weeks after last treatment dose. The women not of reproductive potential are female patients who are postmenopausal (with a minimum of one year without menstruation and without alternative medical cause) or permanently sterilized: e.g., tubal occlusion, hysterectomy, bilateral salpingectomy).
10. Must be geographically accessible for follow-up
11. Written and dated informed consent
12. Affiliated to the French national social security system

Exclusion Criteria:

1. Current treatment by : statin, fibrate, ciclosporin, systemic fusidic acid, long-term treatment by corticoids
2. History of muscular dystrophy diseases or chronic and/or hereditary muscular diseases
3. Patients with distant metastases
4. Indications of node irradiation (axillar or supraclavicular or mammary chain)
5. T3-4 or N1-3 breast cancer
6. Patients who underwent radical mastectomy
7. Neoadjuvant systemic therapy (chemotherapy, hormonotherapy, targeted therapies)
8. Patients with previous or concomitant other (not breast cancer) malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for at least five years
9. Patients with other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung embolism, infection etc.) which would disrupt extended follow-up
10. Untreated hypothyroidism
11. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody
12. Pregnant or breastfeeding women
13. women of childbearing potential who are unwilling to employ adequate contraception, from the beginning of the study to 4 weeks after last treatment dose
14. Known hypersensitivity to pravastatine, or any constituent of the product.
15. Patient with alcohol misuse.
16. Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Impact of Pravastatin on the occurrence of grade ≥2 breast fibrosis in a selected breast cancer patient population considered at high risk of severe breast fibrosis occurrence | From randomization to 24 months
  2-year breast fibrosis-free survival (BF-FS) rate

SECONDARY OUTCOMES:
Impact of this personalized radiotherapy on Acute toxicities | from randomization to 3 months
  Incidence of acute effects assessed and graded according to the NCI-CTCAE v5.0 scale; the most severe grade observed during the period per patient will be reported.
Impact of this personalized radiotherapy on late toxicities | from randomization to 3 years
  late side effects assessed and graded according to the NCI-CTCAE v5.0 scale; the most severe grade observed during the period per patient will be reported.
Adverse events due to Pravastatine | from randomization to 2 years
  rate of myalgia and arthralgia
Local recurrence | at 1, 2, 3, 5 and 10 years
  Local recurrence rate
Relapse free survival (RFS) | at 1, 2, 3, 5 and 10 years
  Relapse-free survival (RFS) rates with RFS defined as the time from the date of randomization to the date of the first relapse (including local relapse, or distant metastasis or death (all causes), whichever occurs first.
Breast fibrosis-free survival (BF-FS) | at 6 months, at 1 and 3 years
  BF-FS rates
Breast fibrosis-relapse-free survival (BF-RFS) | at 1, 2, 3 and 5 years
  BF-RFS rates with BF-RFS defined as the time from the date of randomization to the date of the first relapse (including local relapse, or distant metastasis or death (all causes) or the first documented grade ≥2 breast fibrosis whichever occurs first.
Specific quality of life measure for breast cancer patient | at baseline, 5 weeks after RT and 6, 12, 18, 24 and 36 months , at 4 and 5 years
  EORTC QLQ-C30 questionnaires : minimum value = 1 (no effect) maximum value = 4 (bad effect)
Specific quality of life measure for breast cancer patient | at baseline, 5 weeks after RT and 6, 12, 18, 24 and 36 months , at 4 and 5 years
  QLQ-BR23 questionnaires:minimum value = 1 (no effect) maximum value = 4 (bad effect)
the Cosmetic affect | at baseline, at 12 months and at 2 years of pravastatin/Placebo treatment
  rate of the acute and rate of later side effects with photographics
feasibility of a new production technique for NovaGray RILA Breast® test | at baseline
  test score sensitivity
Stability of the test | at 12 months
  The radiation-induced lymphocyte apoptosis (RILA) assay is the leading candidate as a biological predictor of radiotherapy toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Céline Bourgier, MD, Study Chair — ICM Co. Ltd.
Locations (7):
- France (6):
  - Centre Azuréen de Cancérologie, Mougins, Alpes-Maritimes
  - Clinique Sainte-Anne, Strasbourg, Bas-Rhin
  - Centre Hospitalier de Brive, Brivé, Corrèze
  - Centre Georges-François Leclerc, Dijon, Côte d'Or
  - Icm Val D'Aurelle, Montpellier, Herault
  - Centre Hospitalier Universitaire Lyon Sud, Lyon
- Centre Hospitalier Princesse Grace, Monaco, Monaco